CLINICAL TRIAL: NCT03011905
Title: Rebound Pain at Block Resolution After Operations for Distal Radius Fractures With a Volar Plate in Brachial Plexus Block
Brief Title: Rebound Pain After Operations for Distal Radius Fractures With a Volar Plate in Brachial Plexus Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anne Holmberg, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/599/REK sør-øst C
Record Dates: First submitted 2016-12-21; First posted 2017-01-05 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Brachial Plexus Block; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Acetaminophen; Etoricoxib; Oxycodone; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Single dose of dexamethasone (Dexagalen) 16 mg iv during operation.
  Interventions: Drug: Dexamethasone; Drug: Paracetamol; Drug: EtoriCoxib; Drug: Oxycodone; Drug: Ropivacaine
- Control (Placebo Comparator): Single dose of NaCl, 4 ml, iv during operation.
  Interventions: Drug: NaCl (Control); Drug: Paracetamol; Drug: EtoriCoxib; Drug: Oxycodone; Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexamethasone — 4 ml DexaGalen 4 mg/ml
  Other Names: DexaGalen
  Arms: Dexamethasone
Drug: NaCl (Control) — 4 ml NaCl 9 mg/ml
  Other Names: NaCl
  Arms: Control
Drug: Paracetamol — Premedication and as needed after operation
Drug: EtoriCoxib — Premedication and first 2 postoperative days.
  Other Names: Arcoxia
Drug: Oxycodone — Total of 3 doses of OxyContin postoperatively. OxyNorm as needed.
  Other Names: OxyContin; OxyNorm
Drug: Ropivacaine — In brachial plexus block

SUMMARY:
Many patients have strong pain at brachial plexus block resolution after operations for distal radius fractures with a volar plate. This study investigates if a single dose of dexamethasone in addition to a standard pain regime have an effect on postoperative pain. The primary endpoint is difference in the highest pain score first 24 hours after surgery. The investigators will also look at pain scores and analgesics consumption first few hours after surgery and at different times up to 2 years after surgery.

DETAILED DESCRIPTION:
This double-blind randomized clinical study evaluates pain, analgesic consumption and different measurements of patients satisfaction after operations for distal radius fractures with a volar plate in the day-care surgery unit. All patients will receive paracetamol and etoricoxib as oral premedication. Patients will be operated in infraclavicular brachial plexus block with ropivacaine 7,5 mg/ml. Patients in the intervention group will receive a single dose of 16 mg dexamethasone during the operation. Patients in the control group will receive NaCl iv.

After surgery, iv and oral rapid release oxycodone as needed while in hospital. After discharge (after 2-4 hours), etoricoxib for 2 days, controlled release oxycodone, total of 3 doses. Rapid release oxycodone as needed.

Patients will be followed up by telephone interviews at different times after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture planned for operation with a volar plate
* 0-20 days after trauma
* AO classification A, B, and C
* ASA 1 and 2
* Age 18-65
* BMI 18-35
* Able to communicate in Norwegian

Exclusion Criteria:

* Chronic pain
* Other injuries
* Pregnancy
* Known allergic reactions to medicines used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
Differences between groups in highest pain scores first 24 hours after surgery | 24 hours

SECONDARY OUTCOMES:
Differences in pain scores after 30 min, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours | 30 min, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours
Differences in pain scores after 36 hours, 3 days, 7 days, 6 weeks | 36 hours, 3 days, 7 days, 6 weeks
Differences in pain scores after 6 months and 1 year | 6 months and 1 year
Differences in analgesic consumption | 1 hours, 2 hours, 4 hours, 8 hours, 24 hours, 36 hours, 72 hours, 1 week, 6 weeks, 6 months, 1 year
Differences in block duration | 20 hours
Differences between groups in sedation postoperatively assessed with Likert scale | 30 min, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours, 36 hours, 72 hours
  Likert scale
Differences between groups in sleep quality assessed with Likert scale | 24 hours
  Likert scale
Differences between groups in nausea postoperatively assessed with Likert scale | 30 min, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours, 36 hours, 72 hours
  Likert scale
Differences between groups in vomiting postoperatively assessed with Likert scale | 30 min, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours, 36 hours, 72 hours
  Likert scale
Differences between groups in itching postoperatively assessed with Likert scale | 30 min, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours, 36 hours, 72 hours
  Likert scale
Differences in time to first pain score under 4 after block resolution | 7 days
Differences in side effects | 1 year
Differences in Patient Rated Wrist/Hand Evaluation (PRWHE) scores after 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holmberg, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo Universitetssykehus, Ullevaal, dept of anaesthesiology, legevakten, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmberg A, Hassellund SS, Draegni T, Nordby A, Ottesen FS, Gulestol A, Raeder J. Analgesic effect of intravenous dexamethasone after volar plate surgery for distal radius fracture with brachial plexus block anaesthesia: a prospective, double-blind randomised clinical trial. Anaesthesia. 2020 Nov;75(11):1448-1460. doi: 10.1111/anae.15111. Epub 2020 May 30. PMID 32472958